CLINICAL TRIAL: NCT01888471
Title: Feasibility Study for Identifying a Sero-correlate of Protection Against Invasive Group B Streptococcus Disease in Newborns and Young Infants Aged Less ≤90 Days
Brief Title: Feasibility Study for Identifying Anti Capsular Antibody Protection Against Invasive Group B Streptococcus (GBS) Disease in Newborns of 0-6 Days Age (Early Onset Disease [EOD]) as Well as Among Infants of 7-90 Days Age (Late Onset Disease [LOD])
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 205523; V98_22OB (Other: Novartis)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Streptococcus Agalactiae
Keywords: Streptococcal disease; Feasibility; Infants
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Cases Group (Other): Cases Group will be defined as:
  Maternal subjects identified with invasive GBS disease from the enrolled maternal-newborn dyad Study cohort: Cases will be classified as follows:
  * EOD (Early onset disease): isolation of GBS from the blood or cerebrospinal fluid (CSF) within 0-6 days of birth.
  * LOD (Late onset disease): isolation of GBS from the blood or cerebrospinal fluid (CSF) within 7-90 days of birth.
  Interventions: Procedure: Blood sample; Other: Vaginal swab sample
- Controls Group (Other): Controls will be defined as newborns to mothers, enrolled into the study and identified as colonized by a serotype which is homologous to that of cases, but who do not develop invasive GBS disease.
  Interventions: Procedure: Blood sample; Other: Vaginal swab sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample will be obtained from enrolled mothers at delivery(either immediately before or after delivery) Both original blood sample and cord blood sample will be obtained for serology.
Other: Vaginal swab sample — Vaginal swab will be collected at delivery from a pre-defined subset of enrolled mothers for the identification of controls, for determining GBS maternal colonization status and serotype.

SUMMARY:
The purpose of this study is to evaluate antibody levels against Group B streptococcus in mothers and the risk of developing invasive Group B streptococcus disease in newborns of less than 6 days age as well as infants of age less than 90 days age.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (irrespective of gestational age staging or underlying comorbidities) attending for antenatal care at Chris Hani Baragwanath Academic Hospital (CHBAH) or an allied antenatal clinic and/or delivering at the participating delivery center (CHBAH)
* Subjects aged ≥18 years.
* Able to understand and comply with planned study procedures.
* Provides written informed consent.

Exclusion Criteria:

• Subjects Refusing to consent to study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women (irrespective of gestational age staging or underlying comorbidities) attending for antenatal care at CHBAH or an allied antenatal clinic and/or delivering at the participating delivery center (CHBAH).
Enrollment: 3033 (Actual)
Dates: Start 2013-12-11 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2014-07-14 (Actual)

PRIMARY OUTCOMES:
Proportion (Percentage) of maternal subjects enrolled in the study relative to the number of pregnant women screened. | During routine antenatal visits in the 4 months enrollment period (in antenatal clinics attached to study delivery units or the clinics serving the population delivering at those unit)
  Maternal mothers were excluded at screening if:
  * Age <18 yrs.
  * Not planning to deliver at study center.
  * Did not consent.
Proportion (percentage) of maternal subjects enrolled in ante-natal clinics. | During routine antenatal visits in the 4 months enrollment period(in antenatal clinics attached to study delivery units)
  Percentage of maternal mothers who were not excluded at screening and who were presenting in antenatal clinics.
Proportion (percentage) of maternal subjects enrolled at delivery. | At delivery
  Percentage of maternal mothers who were not excluded at screening and who were enrolled at delivery visit.
Proportion (percentage) of mother-infant dyads enrolled with data available to assess early censorship criteria. | At delivery
  Percentage of mothers who were not excluded at screening and with data available to assess Early censoring criteria for defining the final analysis population:
  * Intravenous intrapartum antibiotics at delivery.
  * Blood transfusion in the 30 days prior to delivery.
  * Infant born with life threatening condition/ congenital malformation.
  * Failure to complete 90 day Follow-Up for potential controls.
  * Non-homologous serotype in case infants and mothers.
Proportion (percentage) of enrolled mother-infant dyads with cord blood collected. | At delivery
  Percentage of maternal mother (who were not excluded at screening) -infants dyads and with cord blood sample obtained for serology.
Proportion (percentage) of enrolled mother-infant dyads with both maternal and cord blood collected. | At delivery
  Percentage of maternal mother (who were not excluded at screening) -infants dyads and with both maternal and cord blood sample obtained for serology.
Proportion (percentage) of mother-infant dyads with complete data on the defined key clinical variables. | Throughout the study, an average of 4 months.
  Percentage of maternal mother (who were not excluded at screening) -infants dyads with defined key clinical variables.
  The key clinical variables have been defined as follows:
  Maternal subjects
  * Smoking during pregnancy,
  * Vaginal douche during pregnancy,
  * Gestational age at enrolment,
  * HIV test completed during routine care,
  * For those with test completed availability of test result and for HIV positive subjects CD4 count and viral load data.
  * Time between rupture of membranes and delivery,
  * Intrapartum antibiotic usage at delivery and duration of treatment
  * Evidence of intra-amniotic uterine infection.
  Infant subjects:
  * Birth weight,
  * Head circumference,
  * Congenital malformation,
  * Completion of 90-day follow-up visit in subset of sub-jects (cases and controls) eligible for this visit.
Percentage of subjects who completed the 90-day follow up visit in subset of subjects eligible for this visit. | At 90 day follow up visit
Percentage of maternal subjects, with vaginal swab samples, culture positive for GBS. | Throughout the study, an average of 4 months.
Percentage of maternal subjects who had culture positive for GBS, classified by serotype. | Throughout the study, an average of 4 months.
GBS anti-capsular antibody concentration (serotype-specific anti capsular antibody) in maternal subjects, vaginally colonized with GBS. | At delivery
GBS anti-capsular antibody concentration (serotype-specific anticapsular antibody) in infant subjects. | At birth

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cutland CL, Cunnington M, Olugbosi M, Jones SA, Hugo A, Maharaj K, Slobod K, Madhi SA. Lessons learnt from enrolment and follow up of pregnant women and their infants in clinical trials in South Africa, a low-middle income country. Vaccine. 2015 Nov 25;33(47):6406-12. doi: 10.1016/j.vaccine.2015.08.040. Epub 2015 Sep 26. PMID 26409812